CLINICAL TRIAL: NCT01045369
Title: A Phase IV 48 Week, Open Label, Pilot Study of Kaletra and Intelence Tablets in Naive Subjects
Brief Title: A Pilot Study of Kaletra and Intelence Tablets in Naive Subjects
Acronym: KALYINTE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Therapeutic Concepts (Other)
Collaborators: Abbott (Industry); Tibotec, Inc (Industry); BluKyne (Unknown)
Responsible Party: Principal Investigator, Joseph Gathe Jr. M.D., MD, Therapeutic Concepts
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 101-001
Record Dates: First submitted 2010-01-08; First posted 2010-01-11 (Estimated); Last update posted 2017-05-01 (Actual); Status verified 2010-01

CONDITIONS: HIV Infections
Keywords: HIV; Treatment Naive
MeSH Terms: conditions — HIV Infections | interventions — lopinavir-ritonavir drug combination; etravirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Kaletra And Intelence (Experimental): This is a Phase IV, 48-week, open-label, pilot study in 30 ARV-naïve patients examining the safety, viral response, and tolerability of Kaletra® and Intelence™ tablets.
  Interventions: Drug: Kaletra and Intelence Tablets

INTERVENTIONS:
Drug: Kaletra and Intelence Tablets — Kaletra 400 mg twice a day and Intelence Tablets 200mg twice a day.

SUMMARY:
The purpose of this study is to see if using a combination of other drug classes, like the ones that Kaletra® and Intelence™ belong to, can still help reduce the amount of HIV in your blood. Using Kaletra® and Intelence™ without other drugs is not approved by the FDA and so their use in this study is experimental.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 RNA ≥ 5000 copies/mL by Roche Amplicor 1.5v Primer
* More than 18 years of age
* Provide written informed consent and willingness to participate in and comply
* Less than 7 days of prior ART with any licensed or investigational compound
* Does not currently have or has not been treated for an active opportunistic infection (OI) within 30 days of screening
* Vital signs, physical examination and laboratory results do not exhibit evidence of acute illness
* A female who is a non-childbearing potentiator or if in child-bearing potential, has a negative serum pregnancy test at screen and agrees to one of the following: complete abstinence from intercourse from 2 weeks prior to administration of the study drug, throughout the study, and for at least 2 weeks after completion or premature discontinuation from the study to account for elimination of the investigational drug. Should a patient decide to become sexually active during the course of the study, she must be counseled and be willing to use one of the birth control methods like double barrier method, intrauterine device, sterilization and any other methods.

NOTE: Data are insufficient to exclude a clinically important interaction of LPV/r with drugs, such as hormonal contraceptives, that are highly metabolized by the cytochrome P450 enzyme system. As a result, hormonal contraception is not considered adequate.

Exclusion Criteria:

* Patient with active AIDS-defining opportunistic infection in the 30 days prior to baseline and that, in the opinion of the investigator, would preclude the patient from participating in the study (See Appendix C).
* Patient has a weighted genotypic score for etravirine ≥3 . (See Appendix D)
* Patient has >3 mutations at 10, 20, 24, 32, 33, 36, 46, 47, 48, 50, 54, 73, 82, 84, or 90 in protease or ≥1 of the following mutations in protease (I47A/V, V32I, or L76V).
* History of active substance abuse.
* Pregnant at time of screening evaluation or breast-feeding.
* Patient, in the opinion of the investigator, is unlikely to be able to complete the 48-week dosing period and protocol evaluations and assessments or adhere to the study drug regimen.
* Serious medical condition, such as diabetes, congestive heart failure, cardiomyopathy or other cardiac dysfunction, which in the opinion of the investigator would compromise the safety of the patient
* Malabsorption syndrome or other gastrointestinal dysfunction, which may interfere with drug absorption or render the patient unable to take oral medication.
* Undergoing interferon therapy for HCV or anticipates undergoing therapy during the course of this trial
* HBV co-infection
* Laboratory results within 30 days prior to the first dose of study medication:

  * Hemoglobin concentration < 8.0 g/dL
  * Absolute neutrophil count < 750 cells/mm3
  * Platelet count <50,000 cells/ mm3
  * Aminotransferase (AST, ALT) >3 times ULN
  * Serum creatinine >1.5 times the Upper Limits of Normal (ULN)
* Radiation therapy or cytotoxic chemotherapeutic agents within 4 weeks prior to entry, or has an anticipated need for these agents within the study period.
* Immunomodulating agents, such as systemic corticosteroids, interleukins, or interferon's within 4 weeks prior to study entry, or patients who have received an HIV immunotherapeutic vaccine within 3 months prior to entry. Asthmatic patients using inhaled corticosteroids are eligible for enrollment.
* Methadone therapy
* Foscarnet therapy or therapy with other agents with documented activity against HIV-1 in vitro.
* Taking astemizole, terfenadine, cisapride, oral midazolam, triazolam, flecainide, pimozide, propafenone, St. John's Wort, lovastatin, simvastatin, and rifampin or ergot derivatives.
* Allergy to any of the study drugs or any excipients therein.
* Patient requires inhaled or intranasal fluticasone.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-04 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with plasma HIV-1 RNA < 400 copies/mL at weeks 24 and 48 | At weeks 24 and 48
Proportion of patients with plasma HIV-1 RNA < 75 copies/mL at weeks 24 and 48 | At weeks 24 and 48

SECONDARY OUTCOMES:
Proportion of patients with plasma HIV-1 RNA < 400 copies/mL or < 75 copies/mL at each study visit | At weeks 24 and 48
Number of weeks until HIV RNA < 400 copies/mL and < 75 copies/mL, respectively | At weeks 24 and 48

CONTACTS AND LOCATIONS:
Overall Officials: Joseph C. Gathe, Jr., MD, Principal Investigator — Therapeutic Concepts
Locations (1):
- Therapeutic Concepts, PA, Houston, Texas, United States